CLINICAL TRIAL: NCT00968734
Title: Vitamin D Status After Single Oral Dose of Cholecalciferol in Low Fat Meal Compared to High-fat Meal
Acronym: VITDAB_08606
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Fabiana Viegas Raimundo, Universidade Federal do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FIPE, CAPES; GPPG_080606
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2009-08

CONDITIONS: Deficiency, Vitamin D
Keywords: Vitamin D; colecalciferol; absorption by Vitamin D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low fat meal (Experimental)
  Interventions: Dietary Supplement: colecalciferol
- Hight fat meal (Experimental)
  Interventions: Dietary Supplement: colecalciferol

INTERVENTIONS:
Dietary Supplement: colecalciferol — 50.000UI single oral dose

SUMMARY:
The purpose of this study is to evaluate the absorption of dietary supplement of vitamin D3 (cholecalciferol), through the variation of 25 (OH) D levels, as the fat content of the meal associated with the administration of the supplement.

DETAILED DESCRIPTION:
Clinical randomized controlled double-blind study with healthy subjects to investigate the effect of low and high fat of meal on absorption of vitamin D supplement. Participants were randomly in two groups according to sex and BMI.

In the same date, each group of participants received a meal and dietary supplement of vitamin D3 (cholecalciferol) after the first blood sample and a urine sample. Others samples were collected in the seventh and fourteenth day after intake the supplement.

ELIGIBILITY:
Inclusion Criteria:

* Residents of the hospital clinics of Porto Alegre

Exclusion Criteria:

* Don't drink milk
* Obesity
* Malnutrition
* Liver disease
* Kidney disease or diabetes
* Use of dietary supplements containing calcium and vitamin D
* Medications
* Anticonvulsants
* Barbiturates, or steroids.
* Having performed a journey the last four months to locations near the Earth's equatorial plane, due to sun exposure that may have occurred during this period, or vacations planned during the study period.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Serum Level of Vitamin D3 | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana Viegas Raimundo, graduation, Principal Investigator — Federal University of Rio Grande do Sul; Tania Weber Furlanetto, PhD, Study Director — Federal University of Rio Grande do Sul; Gustavo Faulhaber, Master, Principal Investigator — Federal University of Rio Grande do Sul; Rosana Scalco, Master, Principal Investigator — Hospital de Clínicas de Porto Alegre; Leonardo Marques, Graduation, Principal Investigator — Hospital de Clínicas de Porto Alegre; Paula Menegatti, Graduation, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil